CLINICAL TRIAL: NCT07039630
Title: A Sustainable Nutrition Security Intervention for Low-Income Households
Brief Title: A Food Security Intervention for the Prevention of Cancer in Low-income Families
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: behavioral intervention is being prepared
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: UB Clinical and Translational Science Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IC-4480925; NCI-2025-03869 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IC-4480925 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-06-10; First posted 2025-06-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Obesity-Related Malignant Neoplasm
MeSH Terms: interventions — Food Assistance; Health Promotion; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (enhanced food box, educational materials, call) (Experimental): Participants receive enhanced delivery half-price food boxes delivered by a community health worker and assistance on the proper handling and storage of the food over 24 weeks on study. Participants receive nutritional education materials and access to additional educational resources on the FreshFix online ordering platform. Participants also receive a dietary recall phone call at baseline and at 6 months on study.
  Interventions: Behavioral: Food Assistance Programs; Other: Health Promotion and Education; Other: Questionnaire Administration; Other: Survey Administration; Behavioral: Telephone-Based Intervention
- Arm II (standard food box) (Active Comparator): Participants receive the standard half-price produce box delivery delivered by FreshFix staff over 24 weeks on study.
  Interventions: Behavioral: Food Assistance Programs; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Behavioral: Food Assistance Programs — Receive enhanced delivery half-price food boxes delivered by a community health worker
  Arms: Arm I (enhanced food box, educational materials, call)
Behavioral: Food Assistance Programs — Receive the standard half-price produce box delivery delivered by FreshFix staff
  Arms: Arm II (standard food box)
Other: Health Promotion and Education — Receive nutritional education materials and resources
  Arms: Arm I (enhanced food box, educational materials, call)
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies
Behavioral: Telephone-Based Intervention — Receive a dietary recall phone call
  Arms: Arm I (enhanced food box, educational materials, call)

SUMMARY:
This study is being done to see how produce delivery with or without nutritional education affects what people eat and if it can help improve diet and nutrition in low-income families and their ability to get enough healthy food. Research shows strong evidence regarding the role of diet in new cancer rates and cancer deaths. Although dietary guidelines have been established at the national level to improve diet quality, the average dietary quality remains low in American households, particularly in low-income communities. These disadvantaged communities are also more likely to be food insecure (having limited or uncertain access to nutritious food). FreshFix is a community-based organization that provides nutritious foods from local farmers to communities in Western New York and offers a Half-Price Produce delivery program which is targeted for lower-income and underserved communities. Participating in the FreshFix program with access to nutritional education materials may decrease food insecurity and improve diet quality in low-income families.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop a nutrition security intervention to improve the nutrition security of low-income households.

II. To determine the feasibility of the nutrition security intervention.

SECONDARY OBJECTIVE:

I. To refine the intervention by engaging community-based organizations and households enrolled in the nutrition security intervention to ascertain the barriers and facilitators of intervention implementation.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive enhanced delivery half-price food boxes delivered by a community health worker and assistance on the proper handling and storage of the food over 24 weeks on study. Participants receive nutritional education materials and access to additional educational resources on the FreshFix online ordering platform. Participants also receive a dietary recall phone call at baseline and at 6 months on study.

ARM II: Participants receive the standard half-price produce box delivery delivered by FreshFix staff over 24 weeks on study.

ELIGIBILITY:
Inclusion Criteria:

* Lives in Western New York (WNY)
* Is the person responsible for at least half of the food purchasing and preparation
* Categorized as having marginal, low of very low food security
* Able to access to internet and e-mail/text messages
* Speaks and understands English

Exclusion Criteria:

* Participants that are unable to speak and understand English
* Participants that are unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant(s) is/are an unsuitable candidate to receive the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in nutrition security | Baseline to 24 weeks
  Diet quality will be assessed by recall interview administered through the Nutrition Data System for Research.
Intervention acceptability | At 24 weeks
  Conducted at 24 week follow up via phone or text based survey

CONTACTS AND LOCATIONS:
Overall Officials: Karen Yeary, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States